CLINICAL TRIAL: NCT06047106
Title: DOVIMIR : Multi-parametric MRI Evaluation of Renal Graft Performance After Living Donor Donation
Brief Title: Multi-parametric MRI Evaluation of Renal Graft Performance After Living Donor Donation.
Acronym: DOVIMIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_0324; 2023-A01402-43 (Other: ID-RCB)
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Living Donor Donation; multiparametric MRI; ischemia reperfusion injury; kidney graft
MeSH Terms: conditions — Renal Insufficiency, Chronic; Reperfusion Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Monocentric, Prospective, Non-randomized, Exploratory Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living kidney donor (Experimental): Patient eligible for living kidney donation with eGFR > 60 ml/min/1.73m²
  Interventions: Radiation: multiparametric MRI; Biological: blood samples; Biological: urine specimens
- Recipient of kidney transplant from living donor (Experimental): Patient with end-stage chronic kidney failure awaiting kidney transplant from living donor
  Interventions: Radiation: multiparametric MRI; Procedure: kidney graft biopsy; Biological: blood samples; Biological: urine specimens

INTERVENTIONS:
Radiation: multiparametric MRI — For the living donor, multiparametric MRI will be added in the day hospital: at the pre-transplant assessment and at the 12-month post-transplant assessment.
  For the recipient: multiparametric MRI will be added in the day hospital at the time of the systematic assessment at 1 month post-transplant, and will be added in the day hospital at the time of the 12-month post-transplant assessment.
Procedure: kidney graft biopsy — Biopsy of the graft itself prior to transplantation in the recipient.
  Arms: Recipient of kidney transplant from living donor
Biological: blood samples — For donors who are not selected to donate their kidney, a total of 4 mL of blood will be collected at inclusion.
  For donors eligible to donate, a total of 8 mL of blood will be collected (at inclusion and at 12 months post-transplant).
  For recipients, a total of 32 mL of blood will be collected (pre-transplant, 1 month and 12 months post-transplant).
Biological: urine specimens — For donors who are not selected to donate their kidney, a total of 15 mL of urine will be collected at inclusion.
  For donors eligible to donate, a total of 50 mL of urine will be collected (at inclusion and at 12 months post-transplant).
  For recipients, a total of 65 mL of urine will be collected (pre-transplant, 1 month and 12 months post-transplant).

SUMMARY:
The selection of kidneys from living donors is based on strict glomerular filtration rate (GFR) values, in the setting of the increasing proportion of older donors. The 2017 KDIGO recommendations consider that approving kidney donation for a donor with a GFR between 60 and 89 mL/min/1.73 m² should be individually discussed, possibly using a calculator. A GFR < 60 mL/min/1.73 m² should contraindicate donation without considering the donor's age.

GFR physiologically decreases with age, so older donors frequently have a GFR below 90 ml/min/1.73 m². However, the proportion of older donors continues to rise.

Kidney grafts from older living donors maintain better renal function than those from deceased donors, aiming to counteract the organ shortage.

Kidneys possess functional reserves, allowing an increase in GFR during stimulations and adaptation to reduced functional nephron count (as after nephrectomy). Assessing this adaptive capacity clinically is challenging. It might be dependent on vascularization and/or absence of fibrosis, but these parameters are poorly understood due to a lack of current in vivo exploration methods.

The development of functional renal MRI enables the evaluation of these parameters, allowing measurements on separate, regional, non-invasive, quantitative kidney segments coupled with morphological studies. BOLD-MRI can measure regional oxygen content, thus accessing more precise medullary data. The DWI sequence can estimate renal microstructure and study interstitial fibrosis.

Therefore, evaluating renal performance (by measuring GFR, renal perfusion, fibrosis, inflammation, and oxygen content) in donors, and studying the evolution of these parameters in recipients and donors, could optimize donor selection.

Hence, the aim of our study is to 1) investigate the evolution of renal functional parameters in the transplanted kidney up to 1 year post-transplant, and 2) study the evolution of these same parameters in the contralateral kidney of the donor.

ELIGIBILITY:
Inclusion Criteria:

For recipients:

* Patients with end-stage chronic kidney disease awaiting kidney transplant from a living donor.
* Adult patient
* Consent signed
* effective contraceptive method for women
* Patient affiliated to a social security or beneficiaries of a similar scheme

For donors:

* Individuals eligible for living kidney donation with GFR > 60 mL/min/1.73 m².
* Adult patient
* Consent signed
* effective contraceptive method for women
* Patient affiliated to a social security or beneficiaries of a similar scheme

Exclusion Criteria:

For the two groups :

* MRI contraindications (claustrophobia, pacemaker, cardioverter defibrillators implantable, mechanical heart valve non MRI-compatible)
* Weight> 130 kg
* Pregnant, parturient or breastfeeding
* Persons deprived of their liberty by a judicial or administrative decision,
* Adults subject to a legal protection measure (safeguard measure, guardianship, curators)
* subject participating in another research including an exclusion period still in progress at inclusion

For recipients :

- Contraindication to renal graft biopsy (ongoing or uninterrupted anticoagulant or antiplatelet treatment, thrombocytopenia <100 x 10^9/L, anemia <7 g/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Apparent diffusion coefficient (ADC) coefficient values measured in diffusion-weighted MRI sequence | Baseline before transplantation, one month and 12 months after kidney transplantation

SECONDARY OUTCOMES:
In recipients, R2* values measured by BOLD MRI | Baseline before transplantation, one month and 12 months after kidney transplantation
In recipients, T2 Values measured by T2 mapping MRI | Baseline before transplantation, one month and 12 months after kidney transplantation
In recipients, T1 Values measured by T1 mapping MRI | Baseline before transplantation, one month and 12 months after kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine LEMOINE, PU-PH, Principal Investigator — Service de néphrologie à l'Hôpital Edouard Herriot
Locations (1):
- Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon, LYON, France

IPD SHARING:
Plan to Share IPD: No